CLINICAL TRIAL: NCT00747747
Title: Safety and Efficacy (for Symptoms Remission) of the Treatment of the Acute Episode of Sinusitis With Ecballium Elaterium (SINUclean DM® Nasal Spray) as Co-adjuvant of the Antibiotic Therapy: Comparative, Prospective, Randomized, Open Study.
Brief Title: Sinuclean's Treatment Of Sinusitis' Symptoms
Acronym: SToSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galsor S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAL-01-2007; EudraCT: 2007-003739-22 (Other: Sponsor Galsor srl)
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Results first posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Sinusitis
Keywords: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No coadiuvant treatment. The subject is treated with the antibiotic only and forbidden to take any coadiuvant medicine as a remedy for the symptoms during the period of the study.
- Saline solution (Active Comparator): Saline solution sprayed according to the product indication. Only one brand/specific product has been selected.
  Interventions: Biological: Saline solution
- Sinuclean treatment (Experimental): Sinuclean DM Spray.
  Interventions: Device: Sinuclean DM Spray

INTERVENTIONS:
Biological: Saline solution — 3 sprays per nostrils twice a day (morning and evening); in case of need a third nebulization between the two is allowed
  Other Names: Libenar
  Arms: Saline solution
Device: Sinuclean DM Spray — 3 sprays per nostrils twice a day (morning and evening); in case of need a third nebulization between the two is allowed
  Other Names: Sinuclean DM Nasal Spray
  Arms: Sinuclean treatment

SUMMARY:
The goal of the study is to demonstrate that SINUclean DM® spray, added to the standard (amoxicillin/clavulanate) therapy of the acute episode of sinusitis (acute, subacute or chronic), is safe ad capable to determine the resolution of the symptoms in a shorter time in comparison with the standard therapy without co-adjuvant, or with simple saline lavage.

DETAILED DESCRIPTION:
The randomized subject with diagnosis of acute episode of sinusitis with symptoms and mucus in the paranasal sinuses, will treat his/her condition with background amoxicillin/clavulanate and with inhalation of Sinuclean or Saline, while the control group will not use any spray for symptom relief. Anti-histaminic, steroidal anti-inflammatory drugs are forbidden. The patient is requested to evaluate his state of symptoms by recording in a diary

* the pain or feeling of facial oppression;
* nasal dripping anterior or posterior;
* nasal congestion. SCALE 0 = no symptom

  1. = mild symptom: clearly perceptible, but easily tolerated
  2. = moderate symptom: clear awareness of the symptom, that is annoying but tolerable
  3. = severe: symptom very annoying, difficult to tolerate, interfering with the ordinary life Four measures per day (2 for administration of the therapy - before/after) of which the median will be used; plus an evening measure "retrospective" of the past 12 hours.

If possible it will be assessed the status of paranasal sinuses before and after the treatment with a CT scan.

The treatment intervals is the week. After baseline and start of treatment, are planned two control visit. The subject will complete the study at the first control visit without symptoms. After the second visit, if the symptoms are still present, the subject will complete as a "treatment-failure".

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex.
* Age > 18 years old.
* Diagnosis of acute episode of sinusitis (in an acute, subacute or chronic background), confirmed with a CT scan image.
* Presence of mucus in para-nasal sinuses.
* Symptoms of facial pain associated to the congestion of the mucosa of the paranasal sinuses for at least three days.
* Written informed consent.
* Expressed intention of compliance with the study requirements.

Exclusion Criteria:

* In case of female subject: ongoing pregnancy or lactating; or condition of fecundity without abstinence.
* Assumption, during the study, of drugs that can interfere with the evaluation of the investigational drug (see Section "Concomitant Therapy")
* Possible necessity of treatment, during the study, with drugs that are not allowed (see section "Concomitant Therapy").
* Clinical conditions (systemic pathologies or other) that can interfere with the assessment of the safety and efficacy of the investigational drug, in example: viral or allergic rhinitis with active secretive symptomatology, presence of visible nasal polyps, diagnosis of immobile cilia syndrome, diseases determining immunodeficiency cystic fibrosis immunocompromission renal insufficiency, dialysis, pathology of other apparatus that, in the opinion of the investigator, necessity of a supplementary antibiotic therapy,due to other pathologies, besides the one standard of the sinusitis.
* Psychical conditions not compatible with the participation to the clinical trial.
* Alcohol abuse or other dependencies on stupefacents
* Smoking during the period of the study
* History of intolerance or allergy to the components of SINUclean DM®
* Surgical or medical intervention that can jeopardize the complete performance of the trial, in the 4 wks preceding the administration of the informed consent
* Planning of a surgical or medical intervention that can jeopardize the completion of the trial
* Participation to other clinical trials, ongoing or terminated since less than 30 days before the beginning of the present experiment.
* Preceding randomization in this trial.
* Be component of the investigators' staff or be a relative of a member of the staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Paludetti, MD, Principal Investigator — University Cattolica del Sacro Cuore Roma Italy
Locations (1):
- University Cattolica del Sacro Cuore, Rome, Lazio, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period of recruitment: Nov 2007 - Mar 2009 Location: Outpatients attending medical visits by General Practitioners
Groups:
- Saline Treated.: Saline solution sprayed three times in each nostril, twice a day (morning - evening)
- Sinuclean Treated.: Sinuclean sprayed three times in each nostril, twice a day (morning - evening)
Period: Overall Study
Arm/Group | Control | Saline Treated. | Sinuclean Treated.
Started | 14 | 14 | 21
Completed | 14 (13 with acute episode + 1 with recurrent episode) | 14 (11 with acute episode + 3 with recurrent episode) | 21 (17 with acute episode + 4 with recurrent episode)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Saline Treated. | Sinuclean Treated. | Total
Number analyzed (Participants) | 14 | 14 | 21 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 21 | 49
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (15) | 45 (11) | 48 (13) | 47 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 11 | 24
  Male | 6 | 9 | 10 | 25
Region of Enrollment [Number; unit: participants]
  Italy | 14 | 14 | 21 | 49

OUTCOME MEASURES:

1. Primary Outcome: Presence of Mucus in the Paranasal Sinuses (Outcome Measure Percentage of Patients)
Description: Mucus detection in paranasal sinuses by clinical assessment(Outcome measure Percentage of patients)
Time Frame: After one week
Population: The patients were eligible according to inclusion and exclusion criteria and were compliant with the study requirements.
Measure: Number; unit: percentage of patients
Arm/Group | Control | Saline Treated. | Sinuclean Treated.
Number analyzed (Participants) | 14 | 14 | 21
percentage of patients | 71 | 57 | 33
Statistical Analysis 1: Comparison: Control vs Saline Treated. vs Sinuclean Treated; Null hypothesis: no difference among groups; Test type: Superiority or Other; p < 0.05, Chi-squared; Frequency = 0

2. Secondary Outcome: FACIAL PAIN Daily Retrospective Ranking of Symptoms as Assessed by the Subject
Description: Patient's daily diary retrospective ranked assessment of symptoms (0,1,2,3 with 0 = no symptoms; frequencies of patients with rank "0" were compared as outcome measure between groups
Time Frame: After one week
Population: Eligibility per in/ex criteria and compliance with study requirements and diary completion requirements
Measure: Number; unit: percentage of patients
Arm/Group | Control | Saline Treated. | Sinuclean Treated.
Number analyzed (Participants) | 14 | 14 | 21
percentage of patients | 57 | 43 | 52

3. Secondary Outcome: FACIAL PAIN Daily Retrospective Ranking of Symptoms as Assessed by the Subject
Description: as for outcome 2
Time Frame: After two weeks
Measure: Number; unit: percentage of patients
Arm/Group | Control | Saline Treated. | Sinuclean Treated.
Number analyzed (Participants) | 14 | 14 | 21
percentage of patients | 79 | 93 | 81

4. Primary Outcome: Presence of Mucus in the Paranasal Sinuses (Outcome Measure Percentage of Patients)
Description: Mucus detection in paranasal sinuses by clinical assessment(Outcome Measure Percentage of patients)
Time Frame: After two weeks
Measure: Number; unit: percentage of patients
Arm/Group | Control | Saline Treated. | Sinuclean Treated.
Number analyzed (Participants) | 14 | 14 | 21
percentage of patients | 29 | 29 | 15

5. Secondary Outcome: Recovery of Sinusitis Per Clinical Assessment(Outcome Measure Percentage of Patients)
Description: Clinical assessment of healing of the sinusitis episode(Outcome Measure Percentage of patients healed). Healing was assessed clinically by the physician as recovery of the condition prior to the diagnosis of the episode of sinusitis, without need of medical treatment.
Time Frame: After one week
Population: Eligibility according to in/ex criteria and compliance with study requirements
Measure: Number; unit: percentage of patients
Arm/Group | Control | Saline Treated. | Sinuclean Treated.
Number analyzed (Participants) | 14 | 14 | 21
percentage of patients | 29 | 29 | 52

6. Secondary Outcome: Recovery of Sinusitis Per Clinical Assessment (Outcome Measure Percentage of Patients)
Description: Clinical assessment of healing of the sinusitis episode (Outcome Measure Percentage of patients healed. Healing was assessed clinically by the physician as recovery of the condition prior to the diagnosis of the episode of sinusitis, without need of medical treatment.
Time Frame: After two weeks
Measure: Number; unit: percentage of patients
Arm/Group | Control | Saline Treated. | Sinuclean Treated.
Number analyzed (Participants) | 14 | 14 | 21
percentage of patients | 57 | 64 | 90
Statistical Analysis 1: Comparison: Control vs Saline Treated. vs Sinuclean Treated; Null hypotheis: no difference among the groups; Test type: Superiority or Other; p < 0.05, Chi-squared; Frequency = 0

ADVERSE EVENTS:
Time Frame: The period in which Adverse Events were collected was the period of observation of the patient between the Start and the End of the therapy: two weeks maximum.
Description: A 0 frequency means that no events were reported or observed in all the patients of the group considered.
Arm/Group | Control | Saline Treated. | Sinuclean Treated.
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/21
Other Adverse Events (participants affected / at risk) | 0/14 | 1/14 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=14) | Saline Treated. (N=14) | Sinuclean Treated. (N=21)
Flu syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Clinical diagnosis could not be confirmed before treatment start due to logistics problems to make cranial MRI in due time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No